CLINICAL TRIAL: NCT03500367
Title: Efficacy and Safety of Rapamycin (Sirolimus) in the Treatment of Symptomatic Uterine Fibroids and Leiomyomatosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, zhulan, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPMS201802
Record Dates: First submitted 2018-03-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Uterine Fibroids
Keywords: mammilian target of rapamycin inhibitor; Rapamycin (sirolimus); Treatment; Complications
MeSH Terms: conditions — Leiomyoma | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rapamycin (Experimental): rapamycin, 2 mg a day, orally ,for 3months
  Interventions: Drug: rapamycin

INTERVENTIONS:
Drug: rapamycin — rapamycin, 2 mg a day, orally ,for 3months

SUMMARY:
A prospective non-randomized open label clinical trial to research the efficacy and safety of sirolimus in patients with symptomatic, recurrent uterine fibroids or/and various rare leiomyoma.

DETAILED DESCRIPTION:
Recent studies indicate that mTOR pathway is a specific and sensitive tumor target molecule in uterine fibroids, which can be used as a target molecule for interventional therapy and can provide a new cut-in point for nonoperative treatment. However, the application of mTOR inhibitor (sirolimus) in the treatment of uterine fibroids remains blank. Our study was designed as a prospective non-randomized open label clinical trial to research its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria

1. Patients who suffer from menorrhagia and pressure symptoms and whose pelvic ultrasound or pelvic MRI indicates uterine fibroids; or who has underwent myomectomy but suffer from menorrhagia and pressure symptoms again with pelvic ultrasound or pelvic MRI indicating uterine fibroids; or whose other imageological examinations or established surgical diagnosis indicate various rare types of myomatosis and who expect a drug therapy.
2. Symptoms of uterine fibroids can be confirmed if one or multiple symptoms below exist:

   * MP shows an excessive amount of bleeding during menstruation (>80.0 mL)
   * A subject report shows three excessive amounts of bleeding during menstruation in latest six months
   * A subject report indicates pelvic pressure symptoms/pain that are likely related to uterine fibroids.
3. According to results of medical history, physical examinations, gynecological examinations and laboratory examinations, patients are in a good overall condition (except uterine fibroids).
4. Cervical smears show a normal result or have no clinical significance, where further follow-up is unnecessary. If there's a normal result in the latest six month in the medical record of a subject, the subject can pass the inspection of cervical smears. A HPV test can be applied to subjects with equivocal ASCUS as an auxiliary test. ASCUS subjects who get a negative result of a HPV test can be included into this study.
5. Endometrial biopsy should be conducted to eliminate non-endometrial lesions if necessary.
6. Subjects didn't receive any drug therapy for uterine fibroids three months before the clinical test.
7. Female adults have menstruation (>18 years old) and are not during pregnancy and lactation.
8. Subjects have good organ function and results of their biochemical examinations meet the following conditions:

   * AST≤2.5×the upper limit of normal (ULN),
   * ALT≤2.5×the upper limit of normal (ULN),
   * Serum total bilirubin≤1.5×the upper limit of normal (ULN),
   * Creatinine≤1.5×the upper limit of normal (ULN).
9. Patients have signed the informed consent.

Exclusion Criteria

1. Patients are in a period of pregnancy and lactation (patients delivered, miscarried or breast-feed in three months before the treatment)
2. Patients are allergic to any ingredient of the medicine
3. Patients suffer from a disease requiring immediate blood transfusion
4. Patients suffer from a disease that may impact implementation of the study or explanation of results. This type of diseases includes:

   * Known severe blood coagulation disorders
   * Known anemia that is not caused by HMB
   * Known hemoglobinopathy
   * Patients suffered or suffer from cancer of the uterus, cervical carcinoma, ovarian cancer or breast cancer 5) An ultrasonic examination shows one or multiple ovarian cysts with a diameter >30 mm 6) Ovarian tumors or pelvic mass of unknown origin 7) Known or suspected endometrial polyp >15 mm
5. Alcohol or drug (such as aperient) abuse
6. Undiagnosed abnormal bleeding of the reproductive system.
7. Patients also participate in another clinical medicine study
8. Patients took part in another clinical trial that may influence this study before this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
size of uterus and the myoma | 2 day
  efficacy assessment

SECONDARY OUTCOMES:
hormone levels | 2 day
  ovarian function assessment
menstrual blood volume / haemorrhage | 1 day
  symptom assessment
adverse event | 2 day
  safety assessment
follicular size | 2 day
  safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within twelve months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Fritsch M, Schmidt N, Groticke I, Frisk AL, Keator CS, Koch M, Slayden OD. Application of a Patient Derived Xenograft Model for Predicative Study of Uterine Fibroid Disease. PLoS One. 2015 Nov 20;10(11):e0142429. doi: 10.1371/journal.pone.0142429. eCollection 2015. PMID 26588841
- [Background] Prizant H, Sen A, Light A, Cho SN, DeMayo FJ, Lydon JP, Hammes SR. Uterine-specific loss of Tsc2 leads to myometrial tumors in both the uterus and lungs. Mol Endocrinol. 2013 Sep;27(9):1403-14. doi: 10.1210/me.2013-1059. Epub 2013 Jul 2. PMID 23820898
- [Background] Kashani BN, Centini G, Morelli SS, Weiss G, Petraglia F. Role of Medical Management for Uterine Leiomyomas. Best Pract Res Clin Obstet Gynaecol. 2016 Jul;34:85-103. doi: 10.1016/j.bpobgyn.2015.11.016. Epub 2015 Nov 25. PMID 26796059
- [Background] Suo G, Sadarangani A, Tang W, Cowan BD, Wang JY. Telomerase expression abrogates rapamycin-induced irreversible growth arrest of uterine fibroid smooth muscle cells. Reprod Sci. 2014 Sep;21(9):1161-70. doi: 10.1177/1933719114532839. Epub 2014 Apr 30. PMID 24784716
- [Background] Prizant H, Hammes SR. Minireview: Lymphangioleiomyomatosis (LAM): The "Other" Steroid-Sensitive Cancer. Endocrinology. 2016 Sep;157(9):3374-83. doi: 10.1210/en.2016-1395. Epub 2016 Jul 13. PMID 27409646
- [Derived] Zhang G, Fan R, Yang H, Su H, Yu X, Wang Y, Feng F, Zhu L. Safety and efficacy of sirolimus in recurrent intravenous leiomyomatosis, pulmonary benign metastatic leiomyomatosis, and leiomyomatosis peritonealis disseminata: a pilot study. BMC Med. 2024 Mar 13;22(1):119. doi: 10.1186/s12916-024-03344-9. PMID 38481209
- See also: Xenograft Model for Predicative Study of Uterine Fibroid Disease — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=26588841&query_hl=1
- See also: Medical Management for Uterine Leiomyomas — http://linkinghub.elsevier.com/retrieve/pii/S1521693415002308
- See also: Telomerase expression abrogates rapamycin-induced irreversible growth arrest of uterine fibroid smooth muscle cells — http://journals.sagepub.com/doi/10.1177/1933719114532839

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT03500367/Prot_SAP_000.pdf